CLINICAL TRIAL: NCT03427671
Title: An Open Label, Single Center Study to Evaluate the Safety and Effectiveness of OCL 500 Embolization Microspheres (OCL 500) in Uterine Artery Embolization for the Treatment of Premenopausal Women With Symptomatic Uterine Fibroids
Brief Title: OCL 500 Treatment of Women With Symptomatic Uterine Fibroids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMBiotechnologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCL500-P3-UFE-02
Record Dates: First submitted 2018-02-04; First posted 2018-02-09 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Uterine Fibroid; Myoma; Leiomyoma
MeSH Terms: conditions — Leiomyoma; Myoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Occlusin 500 microspheres (Experimental): Uterine fibroid embolization
  Interventions: Device: Occlusin 500 Microspheres

INTERVENTIONS:
Device: Occlusin 500 Microspheres — Occlusin 500 microspheres will be administered using a catheter directed to the uterine vasculature using fluoroscopy. The microsphere suspension will be administered to a near-stasis endpoint.

SUMMARY:
This is a prospective, open-label, single-arm, safety and effectiveness study of Occlusin 500 microspheres in women with symptomatic uterine fibroids.

DETAILED DESCRIPTION:
Prior to entering the study, all patients will undergo pre-study assessments including compliance with inclusion and exclusion criteria, laboratory assessments, pelvic examination, and imaging of the pelvis. Following conventional catheter angiography to confirm catheter placement and the uterine vasculature, each patient will undergo transarterial embolization with Occlusin 500 microspheres.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women with symptomatic uterine fibroids
* Willing and able to provide informed consent
* Fibroids visible by ultrasound or non-contrast magnetic resonance imaging
* Fibroids with a minimum diameter of 4cm for a single fibroid or 3cm where there are 2 or more fibroids; minimum total fibroid burden 33cc
* Documented ovulation by Luteinizing Hormone (LH) testing
* Follicle Stimulating Hormone (FSH) value >40 IU/L within 3 months prior to procedure
* Pelvic examination within 6 months prior to procedure
* Normal Pap smear

Exclusion Criteria:

* Positive pregnancy test
* Uterine size > 20 weeks gestation
* Fibroids that are more than 50% submucosal
* Individual fibroids > 12cm in diameter, or total fibroid burden > 905cc
* Pedunculated subserosal fibroids with an attachment to the uterus less than 50% of the greatest diameter of the fibroid
* Fibroids situated in the cervix
* Abnormally large ovarian arteries
* Uterine pathology other than fibroids
* History of gynecologic malignancy
* Active pelvic infection or history of pelvic inflammatory disease
* Undiagnosed pelvic mass outside the uterus
* History of chemotherapy or radiation to the abdomen or pelvis
* Intra-Uterine Device (IUD) in position
* History of, or ongoing, hemolytic anemia
* Severe cerebrovascular disease defined by a cerebrovascular accident within 6 months of treatment
* Anticoagulant therapy or known bleeding disorder
* Treatment with Gonadotropin Releasing Hormone (GnRH) agonists within the previous 6 weeks
* Received another investigational agent within past 12 weeks
* Compromised hematopoietic function
* Compromised hepatic function
* Compromised renal function
* BMI > 38
* Claustrophobia
* Contraindication to angiography
* Contraindication to magnetic resonance imaging (MRI) or MRI contrast agents
* Allergy to contrast agents
* Allergy to bovine collagen
* Patient desires to become pregnant, or does not agree to contraception during study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Fibroid volume | 6 months post-embolization
  Magnetic Resonance Imaging-determined fibroid volume

SECONDARY OUTCOMES:
Uterine volume | 1 month post-embolization
  Magnetic Resonance Imaging-determined uterine volume
Uterine volume | 6 months post-embolization
  Magnetic Resonance Imaging-determined uterine volume
Fibroid volume | 1 month post-embolization
  Magnetic Resonance Imaging-determined fibroid volume
Quality of Life Assessment | 1 month post-embolization
  Uterine Fibroid Symptom Assessment by Questionnaire
Quality of Life Assessment | 6 month post-embolization
  Uterine Fibroid Symptom Assessment by Questionnaire

OTHER OUTCOMES:
Ultrasound of Uterus | 1 day post-embolization
  Qualitative assessment of uterus comparing baseline to post-embolization time points
Ultrasound of Uterus | 1 month post-embolization
  Qualitative assessment of uterus comparing baseline to post-embolization time points
Ultrasound of Uterus | 6 months post-embolization
  Qualitative assessment of uterus comparing baseline to post-embolization time points

CONTACTS AND LOCATIONS:
Overall Officials: Richard Owen, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No